CLINICAL TRIAL: NCT03609164
Title: Does the Arthroscopic Suture-spanning Augmentation of Single-row Repair in Massive Rotator Cuff Tear Reduce the Retear Rate?
Brief Title: Does the Suture-spanning Augmentation of Single-row Repair in Massive Rotator Cuff Tear Reduce the Retear Rate?
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Taipei Veterans General Hospital, Taiwan (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 104-2314-B-075-082
Record Dates: First submitted 2018-07-17; First posted 2018-08-01 (Actual); Last update posted 2018-08-01 (Actual); Status verified 2018-07

CONDITIONS: Rotator Cuff Tear
Keywords: arthroscopic surgery; massive rotator cuff repair; single-row repair; suture-spanning augmentation
MeSH Terms: conditions — Rotator Cuff Injuries

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Suture-spanning augmentation of single-row repair (Experimental)
  Interventions: Procedure: Suture-bridge augmentation of single-row repair
- single-row repair (Active Comparator)
  Interventions: Procedure: Suture-bridge augmentation of single-row repair

INTERVENTIONS:
Procedure: Suture-bridge augmentation of single-row repair

SUMMARY:
There are several associated structural changes when dealing with massive rotator cuff repair, which include tendon retraction and fragility, muscle atrophy and fatty infiltration, as well as osteoporosis over the tendon insertion. Those changes may lead to difficult in applying double-row repair, suture cutting through the tendon, too much tension over the repair and loosening or pull-out of anchors, which may results in poor tendon-bone healing and subsequent high re-tear rate. Therefore decreasing the tension over the repair site may increase the healing over tendon bone junction as well as decrease the risk of anchors loosening. A suture-spanning augmentation with two set of suture loops passing over musculotendinous junction medially and fixed with anchor at the lateral cortical wall may solve the problem. In order to define the clinical benefit of this adjuvant procedure, a prospective randomized control study is designed to compare the adjunctive reinforce suture with the single-row simple suture repair in massive rotator cuff tear.

Around sixty patients were randomized divided into two groups. The study group was used adjunctive reinforce suture repair technique, which was one lateral cortical anchor holding 2 separated set of transverse looping sutures over the medial musculotendinous junction in addition to single row repair, while the control group was used single row repair technique in simple stitch fashion. All patients will have clinical evaluation in pain (VAS score) and functional recovery (ASES and UCLA score) as well as MRI image for the tendon integrity.

If the suture-spanning augmentation of single-row repair can yield an improved healing rate and fewer complications, massive rotator cuff tear should be repaired earlier in order to prevent the late development of irreparable tear.

ELIGIBILITY:
Inclusion Criteria:

* the pre-operative image (MRI) showing the massive rotator cuff tear (fulfilling one of the following definition a tear with a diameter of 5 cm or more; a complete tear of two or more tendons; one with a coronal length and sagittal width greater than or equal to 2 cm)
* patient was willing and able to provide scores for the study

Exclusion Criteria:

* irreparable rotator cuff tear which was identified pre-operatively or intra-operatively
* glenohumeral or acromioclavicular joint osteoarthritis
* stage III or more of the fatty degenerative of supraspinatus in Goutallier classification
* revision surgery
* patients with bacteremia, a systemic infection, or an infection at the surgical site
* patients who previously attempted or failed a treatment program

Ages: 40 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2015-05-01 (Actual); Primary Completion 2016-04-30 (Actual); Study Completion 2018-06-30 (Actual)

PRIMARY OUTCOMES:
Retear rate | 6 months
  Using MR imaging to determine the presence or absence of rotator cuff retears

SECONDARY OUTCOMES:
Visual Analog Score (VAS) | 2 years
  Record the VAS (pain level from 0-10) by the questionnaire, pre-op/post-op 2-year
The American Shoulder and Elbow Surgeons (ASES) Shoulder Score | 2 years
  Record the ASES score by the questionnaire, focus on joint pain, instability, and activities of daily living, pre-op/post-op 2year
University of California at Los Angeles Shoulder Score (UCLA Shoulder Score) | 2 years
  Record the UCLA shoulder score by the questionnaire, focusing on five sub-scales made up of: active forward elevation and strength (physician reported), pain, satisfaction, and function (patient reported), pre-op/post-op 2-year
Shoulder constant score | 2 years
  Record the shoulder constant score by the questionnaire, focusing on ROM, functional assessment, strength measure, pre-op/post-op 2-year

CONTACTS AND LOCATIONS:
Overall Officials: Hsiao-Li Ma, MD, Study Director — Taipei Veterans General Hospital, Taiwan
Locations (1):
- Hsiao-Li, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Ma HH, Chen KH, Chiang ER, Chou TA, Ma HL. Does Arthroscopic Suture-Spanning Augmentation of Single-Row Repair Reduce the Retear Rate of Massive Rotator Cuff Tear? Am J Sports Med. 2019 May;47(6):1420-1426. doi: 10.1177/0363546519836419. Epub 2019 Apr 18. PMID 30998402